CLINICAL TRIAL: NCT06724835
Title: A Single-center, Single-arm, Dose-escalation Exploratory Clinical Trial of the Safety, Efficacy, and Pharmacokinetics of XKDCT293 (Nectin-4-CAR-T) in Nectin-4-positive Advanced Breast Cancer
Brief Title: Treating Nectin-4-positive Advanced Breast Cancer with XKDCT293 (Nectin-4-CAR-T)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Celconta Life Science Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023YP31H01
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-03

CONDITIONS: Advanced Breast Cancer
Keywords: Nectin-4 positive advanced breast cancer
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: Model Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous targeted Nectin4 chimeric antigen receptor T cell injection (Experimental): Autologous targeted Nectin4 chimeric antigen receptor T cell injection
  Interventions: Drug: XKDCT293; Other: CAR-T cell

INTERVENTIONS:
Drug: XKDCT293 — Autologous targeted Nectin4 chimeric antigen receptor T cell injection
Other: CAR-T cell — Nectin-4-CAR-T

SUMMARY:
A single-center, single-arm, dose-escalation exploratory clinical trial of the safety, efficacy, and pharmacokinetics of XKDCT 293 (Nectin-4-CAR-T) in Nectin-4-positive advanced breast cancer

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label, single-dose dose-finding study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy characteristics of XKDCT 293 (Nectin-4-CAR-T) cell preparation in subjects with Nectin-4-positive advanced breast cancer.

The study will enroll subjects with pathologically confirmed advanced breast cancer, positive Nectin-4 expression, who have previously received standard treatment, failed treatment or cannot tolerate it. Imaging examinations show evaluable tumor lesions.

The study included screening period, PBMC collection, baseline, lymphocyte pre-depletion chemotherapy , rest evaluation, cell transfusion, hospitalization observation period, routine follow-up period, and long-term follow-up period.

The study set up three dose groups, and adopted the classic 3+3 experimental design for dose escalation.

Main purpose:

(1)the safety and tolerability of XKDCT 293 in the treatment of nectin-4-positive advanced breast cancer

Secondary Purpose:

1. the cellular metabolic kinetics and pharmacodynamics of XKDCT 293 in the treatment of nectin-4 -positive advanced breast cancer ;
2. To preliminarily evaluate the efficacy of XKDCT 293 cell preparations in patients with advanced Nectin-4-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

·You must meet all of the following conditions to be eligible for the group：

1. Understand and voluntarily sign the informed consent form;
2. Age at screening ranged from 18 to 75 years (including the cutoff value), regardless of gender;
3. Locally advanced or metastatic breast cancer that is unresectable as confirmed by histology or cytology, including triple-negative breast cancer, Her-2-positive, and HR-positive breast cancer;
4. Histological or cytological tumor specimens were confirmed by immunohistochemistry to have moderate to high expression of nectin-4 (expression intensity ≥2+ and tumor cell positive rate ≥50%);
5. Patients who have received standard systemic treatment for breast cancer recommended by the Breast Cancer Diagnosis and Treatment Guidelines (2022 Edition) and have had imaging or other objective evidence of disease progression after receiving standard treatment; or patients with refractory breast cancer who cannot tolerate standard treatment or have contraindications to standard treatment, and who have at least one measurable lesion (according to RECIST version 1.1, the long diameter of the measurable lesion on spiral CT scan is ≥10mm or the short diameter of the enlarged lymph node is ≥15mm, see Appendix 1 for RECIST version 1.1); Note: Treatment failure is defined as disease progression during treatment or recurrence after treatment.

   Definition of intolerance : the occurrence of grade ≥ IV hematological toxicity, grade ≥ III non-hematological toxicity, or grade ≥ III damage to major organs such as heart, liver, and kidney during treatment (refer to NCI-CTCAE v5.0 standards), or a comprehensive assessment by the investigator.
6. The expected survival time at enrollment was greater than 12 weeks;
7. During screening, laboratory tests must meet the following requirements:

   * White blood cell count ≥3.0×10^9 /L;
   * Neutrophil count ≥1.5×10^9 /L;
   * Lymphocyte count ≥ 0.5 × 10^9 /L;
   * Hemoglobin ≥90 g/L;
   * Platelet count ≥75×10^9 /L;
   * Serum total bilirubin ≤2.0× upper limit of normal (ULN);
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5× ULN; For patients with liver metastases or primary liver tumor lesions, aspartate aminotransferase and alanine aminotransferase should be ≤5×ULN; for patients with a history of Gilbert syndrome/suspected Gilbert syndrome, total bilirubin (TBIL) should be ≤3×ULN;
   * Creatinine <1.5×ULN and endogenous creatinine clearance ≥50 mL/min (creatinine clearance Cockcroft-Gault method: creatinine clearance for men = [(140-age)×body weight (kg)]/[0.818×creatinine (umol/L)]; creatinine clearance for women = [(140-age)×body weight (kg)×0.85]/[0.818×creatinine (umol/L)]).
8. Good lung function, with basic finger saturation ≥ 95% in indoor air environment;
9. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
10. Female subjects of childbearing age must undergo a serum pregnancy study with negative results at screening and before purging, and be willing to use medically approved highly effective contraceptive methods during the study and for at least 1 year after the last study treatment. Male subjects whose partners are female subjects of childbearing age should undergo surgical sterilization or agree to use effective contraceptive methods during the study and for at least 1 year after the last study treatment, and are prohibited from donating sperm within 1 year.
11. Venous access can be established, and peripheral blood mononuclear cell collection can be performed at the investigator's discretion.

Exclusion Criteria:

·Anyone who has any of the following conditions cannot be selected as a subject：

1. Pregnant or breastfeeding women;
2. Those who have a history of allergy to any component of the cell product ;
3. Suffering from other malignant tumors, except for the following: cured non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, superficial bladder cancer, and other malignant tumors with a disease-free survival period of more than 5 years;
4. Hepatitis B surface antigen (HBsAg) positive; Hepatitis B core antibody (HBcAb) positive, and HBV DNA copy number positive; Hepatitis C antibody (HCV-Ab) positive; Anti-Treponema pallidum antibody (TP-Ab) positive; Human immunodeficiency virus antibody (HIV-Ab) positive; Those who meet any of the following conditions;
5. Previous anti-tumor treatment or clinical trial participation:

   1. Previously received CAR-T therapy or other gene-edited cell therapy;
   2. Participated in other clinical studies within 28 days before reinfusion;
   3. Received local radiotherapy within 7 days or at least 5 half-lives (whichever is longer) before apheresis or small molecule chemotherapy drugs;
   4. Daily use of systemic glucocorticoids ≥ 15 mg within 7 days before apheresis, excluding inhaled corticosteroids;
   5. Previously received Nectin-4 targeted therapy;
6. Live vaccine or live attenuated vaccine received within 4 weeks before single collection;
7. Surgery has been performed within 2 weeks before apheresis and the researchers believe that it may affect the patient's safety;
8. The investigators judged that there were comorbidities that required the use of systemic corticosteroids or other immunosuppressive drugs during the study;
9. Those who are known to have life-threatening hypersensitivity reactions or other intolerances to cyclophosphamide or fludarabine or severe allergic constitutions; those who have hypersensitivity constitutions, are allergic to human serum albumin, DMSO, etc.; those who are allergic to commonly used first aid and anesthetic drugs;
10. Suffering from any unstable circulatory system disease within 180 days prior to screening, including but not limited to unstable angina, myocardial infarction, heart failure [New York Heart Association (NYHA) grade ≥ III], severe arrhythmia requiring medication, or cardiac angioplasty, coronary artery stenting, or heart bypass surgery within 180 days prior to screening;
11. Uncontrolled diabetes (glycosylated hemoglobin>8%), uncontrolled hypertension (systolic blood pressure/diastolic blood pressure>160mmHg/100mmHg while taking medication);
12. Patients with active infection or uncontrollable infection requiring systemic treatment;
13. The presence or history of central nervous system disease, such as epilepsy, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the CNS;
14. Active autoimmune diseases (including but not limited to systemic lupus erythematosus, Sjögren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, Hashimoto's thyroiditis, etc., except for hypothyroidism that can be controlled only by hormone replacement therapy);
15. Bleeding and thrombotic tendency: clinically significant bleeding symptoms or clear bleeding tendency, such as bleeding gastric ulcer, within 90 days before screening; hereditary or acquired bleeding and thrombotic tendency (such as hemophilia, coagulation disorder, hypersplenism, etc.); currently receiving thrombolytic or anticoagulant therapy; arterial/venous thrombotic events within 180 days before screening, such as cerebrovascular disease (including cerebral hemorrhage, cerebral infarction, etc.), deep vein thrombosis and pulmonary embolism, etc.;
16. Acute toxicity caused by previous treatment has not recovered to grade 1 or below (except hematological toxicity, alopecia, and events judged to be tolerable by the investigator);
17. Those who have a history of psychotropic drug abuse and are unable to quit, or those with a history of mental disorders;
18. The researcher believes that the patient is not suitable for this clinical study (e.g., poor compliance, drug abuse, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days of single infusion
  Dose limiting toxicity (DLT) in the dose escalation phase
Incidence of Treatment Related adverse events (AEs) | 1 year
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs)
Maximum tolerated dose (MTD) | 28 days of single infusion
  Maximum tolerated dose (MTD) in the dose escalation phase

SECONDARY OUTCOMES:
Cellular metabolic kinetics indicators | 1 year
  C max of the number of copies of CAR in peripheral blood of XKDCT293 , the time to reach the maximum concentration T max , the area under the curve for 28 days/90 days AUC 28d /AUC 90d and other related PK parameters and the correlation between cytokines and efficacy
objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS) | 1 year
  To evaluate the objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- AnYang Tumor Hospital, Anyang, Henan, China

IPD SHARING:
Plan to Share IPD: No